CLINICAL TRIAL: NCT03277534
Title: Effects of 8-week Sensory Electrical Stimulation Combined With Motor Training on EEG-EMG Coherence and Motor Function in Individuals With Stroke
Brief Title: Electrical Stimulation Combined With Motor Training on EEG-EMG Coherence and Motor Function in Individuals With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Associate professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 104-2314-B-010-024
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Stroke
Keywords: electrical stimulation
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical stimulation (Experimental)
  Interventions: Other: Electrical stimulation
- Control (Sham Comparator)
  Interventions: Other: Sham electrical stimulation

INTERVENTIONS:
Other: Electrical stimulation — sensory electrical stimulation was applied prior to upper limb functional training
  Arms: Electrical stimulation
Other: Sham electrical stimulation — electrodes were placed on the same location as the Electrical stimulation condition, but no electric current was applied
  Arms: Control

SUMMARY:
This study investigated whether electrical stimulation (ES) prior to a hand function training session for a total of eight weeks can better improve neuromuscular control and hand function in subacute stroke individuals and change electroencephalography-electromyography (EEG-EMG) coherence, as compared to the control (sham ES).

DETAILED DESCRIPTION:
Subjects were randomly assigned into ES and control groups. Both groups received 20-minute hand function training twice a week, and the ES group received 40-minute ES on the median nerve of the affected side before each training session. The control group received sham ES - electrodes were placed on the same location but no electric current was applied. EEG, EMG and Fugl-Meyer Assessment (FMA) were collected before, at the 4th week, at the end of 8th week, and 4 weeks after the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. first-ever cerebral cortical region involved chronic stroke, onset over a month,
2. able to perform active thumb flexion on the affected side with the scores of manual muscle test at least two points, and
3. at stable medical condition for intervention

Exclusion Criteria:

1. history of other neurological disorders,
2. cognitive impairment (Mini-Mental State Examination score <24, MMSE),26
3. unable to follow orders,
4. contraindications of ES, and
5. under 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | before intervention, four weeks after, at the end of the eight-week intervention and four weeks after the intervention period ended
  evaluate changes in upper extremity function of the stroke subjects
EEG-EMG coherence | before intervention, four weeks after, at the end of the eight-week intervention and four weeks after the intervention period ended
  evaluate changes in functional connectivity between motor cortex and active muscles